CLINICAL TRIAL: NCT07012109
Title: A Multicenter, Open-Label Phase I Clinical Trial of BEBT-507 Injection in Subjects With Polycythemia Vera (PV)
Brief Title: Study of BEBT-507 Injection in Subjects With Polycythemia Vera (PV)
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: BeBetter Med Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GBMT-507-P01
Record Dates: First submitted 2025-05-29; First posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-05

CONDITIONS: Polycythemia Vera
Keywords: BEBT-507; Safety; Pharmacokinetics; Efficacy
MeSH Terms: conditions — Polycythemia Vera

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phase Ia-Dose Escalation (Experimental): Phase Ia plans to set up 5 dose groups. If no DLT is observed in cohort A5, further dose escalation will be determined by investigators and sponsors based on PK and safety data. Additional dose groups can be added if necessary.
  Interventions: Drug: BEBT-507 Injection
- Phase Ib-Dose Expansion (Experimental): Based on the results of the phase Ia study, two doses will be selected for the phase Ib study.
  Interventions: Drug: BEBT-507 Injection

INTERVENTIONS:
Drug: BEBT-507 Injection — The initial dose of BEBT-507 injection is 1.25mg/kg, administered subcutaneously at 1.25mg/kg, 2.5mg/kg, 5mg/kg, 10mg/kg or 15mg/kg every 12 weeks for two doses in total.

SUMMARY:
This is a multicenter, open-label Phase I clinical trial of BEBT-507 in subjects with polycythemia vera(PV). Phase Ia is a single-agent dose-escalation study designed to evaluate the safety, tolerability, pharmacokinetics (PK), preliminary efficacy, and pharmacodynamics of BEBT-507 in subjects with PV . Based on the results of Phase Ia, two doses will be selected for further evaluation in Phase Ib to assess the efficacy, safety, and PK profile of BEBT-507 in subjects with PV , and to recommend a dose for Phase III clinical trials.

DETAILED DESCRIPTION:
Phase Ia Study:Phase Ia plans to set up 5 dose groups (Cohorts A1-A5), with 3-6 subjects planned for enrollment in each dose group. The 5 dose groups are 1.25 mg/kg, 2.5mg/kg, 5mg/kg, 10mg/kg, and 15mg/kg, respectively. Subcutaneous injection is administered every 12 weeks, for a total of 2 doses. A "3+3" dose-escalation design will be used. If no dose-limiting toxicity (DLT) is observed in Cohort A5, further dose escalation will be determined by investigators and sponsors based on PK and safety data. Additional dose groups can be added if necessary.

Phase Ib Study:Based on the results of the Phase Ia study, two doses will be selected for the phase Ib study. Each dose cohort will enroll approximately 10-30 eligible subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects aged 18-75 years (inclusive);
2. Subjects diagnosed with polycythemia vera (PV) according to the 2016 world health organization (WHO) criteria;
3. Hydroxyurea-resistant/intolerant and/or interferon α-resistant/intolerant:

1)Hydroxyurea-resistant or -intolerant Must meet the definition of hydroxyurea (HU) resistance or intolerance in the 2024 chinese society of clinical oncology (CSCO) Guidelines for the diagnosis and treatment of malignant hematological diseases and satisfy at least one of the following criteria:a) Resistance: Despite ≥3 months of HU treatment at a dose of ≥2 g/d, phlebotomy is still required to maintain HCT <45%; after ≥3 months of HU treatment at a dose of ≥2 g/d, bone marrow proliferation remains uncontrolled (e.g., platelets >400×10⁹/L and WBC >10×10⁹/L); after ≥3 months of HU treatment at a dose of ≥2 g/d, a palpable massive splenomegaly fails to reduce by >50% or splenomegaly-related clinical symptoms do not fully resolve;b) Intolerance: At the minimum hydroxyurea (HU) dose required to achieve a complete or partial clinical hematologic response for the disease, absolute neutrophil count (ANC) <1.0×10⁹/L or PLT count <100×10⁹/L or Hemoglobin (HGB) <100 g/L occurs; during HU treatment at any dose, lower extremity ulcers or other intolerable non-hematological toxicities emerge, such as skin and mucous membrane manifestations (skin, teeth, or nail darkening; oral ulcers, mucositis; skin ulcers, rash, etc.), gastrointestinal symptoms (nausea, anorexia, indigestion, vomiting, abdominal pain, constipation, etc.), pneumonia, fever, etc.; 2)Interferon α-resistant or -intolerant Must satisfy at least one of the following criteria:a) Resistance: After achieving at least 12 weeks of interferon α therapy and a dose of at least 25×10⁶ U/week (or the subject's maximum tolerated dose if it is less than 25×10⁶ U/week), phlebotomy is still required to maintain HCT <45%, or PLT >400×10⁹/L and WBC >10×10⁹/L, or palpable splenomegaly (starting >10 cm from the left costal margin) fails to reduce by >50%;b) Intolerance: At the minimum interferon α dose required for complete or partial clinical hematologic remission, ANC <1.0×10⁹ or PLT <100×10⁹ or hemoglobin <100 g/L (<10 g/dL) occurs, or depression, influenza-like symptoms, neuropsychiatric symptoms, autoimmune issues, or other unacceptable non-hematological toxicities related to interferon-alpha (IFN-α) emerge, defined as common terminology criteria for adverse events (CTCAE) V5.0 grade 3-4 events, or CTCAE V5.0 grade 2 events lasting over 1 week, or permanent discontinuation of interferon α, or interruption of interferon α until toxicity resolves, or hospitalization due to interferon α toxicity.

4.The subject has intact skin at the injection site, and the investigator deems it is suitable for subcutaneous injection; 5.Eastern cooperative oncology group (ECOG) performance status score is 0, 1, or 2; 6.The subject has undergone bone marrow biopsy within 12 months prior to enrollment; 7.The subject or the subject's legal guardian has signed a written informed consent, and the subject is able to comply with the study requirements.

Exclusion Criteria:

1. A history of intolerance to oligonucleotides, N-Acetylgalactosamine (GalNAc), or excipient components, or a history of intolerance to subcutaneous injections.
2. Clinically significant thrombosis (e.g., deep vein thrombosis or splenic vein thrombosis) within 12 weeks before screening.
3. Major bleeding event or blood transfusion for bleeding within 6 months before screening.
4. Meets the international working group for myeloproliferative neoplasms research and treatment criteria for post-PV myelofibrosis.
5. Received any investigational drug within 6 weeks before the first study drug administration, or not recovered from the effects of prior investigational drugs.
6. Received any clinical studies or marketed products of GalNAc-targeted drugs within 48 weeks before the first study drug administration.
7. Laboratory abnormalities:a) Liver function tests: alanine aminotransferase (ALT) or aspartate aminotransferase (AST)>2.0×Upper Limit of Normal (ULN), total bilirubin（TBIL）>1.5×ULN;b) Renal function tests: estimated glomerular filtration rate (eGFR)<60 mL/min/1.73㎡ (Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation);c) Blood routine tests: platelet count>1000×10⁹/L, WBC count>25×10⁹/L;d) Coagulation tests: international normalized ratio (INR)>1.5×ULN;e) Others: presence of peripheral blood blasts.
8. Subjects with symptomatic splenomegaly (e.g., splenic infarction, left upper quadrant fullness or pain, early satiety, portal hypertension).
9. Due to potential genotoxicity, mutagenicity, and teratogenicity of the study drug, exclude:a) Men and women planning to conceive within 5 years without prior in vitro sperm/ovum preservation;b) Pregnant or breastfeeding women;c) Women within 2 years of menopause unwilling to use acceptable contraception until 6 months after the last study drug dose.
10. Presence of other active malignancies requiring treatment that may interfere with the study.
11. Comorbid conditions:a) Poorly controlled diabetes (random glucose≥11.1mmol/L or HbA1c≥8.5% despite antidiabetic treatment) assessed by the investigator;b) Severe pulmonary disease (CTCAE V5.0 grade III-IV);c) Severe cardiac disease (defined as any of the following:Left ventricular ejection fraction (LVEF) <50% as determined by multigated acquisition scan (MUGA) or Echocardiogram (ECHO);QT interval corrected using the Fridericia method (QTcF) interval >450 ms for males or >470 ms for females;Unstable angina;Symptomatic pericarditis;Myocardial infarction within the past 6 months with persistent elevation of cardiac enzymes or evidence of persistent regional wall abnormalities on LVEF assessment;History of congestive heart failure (new york heart association functional class III-IV) or cardiomyopathy;d) Significant renal or hepatic impairment;e) Poorly controlled active hepatitis B or C, or other diseases with clinically significant active infections, including hepatitis B (HBV), hepatitis C (HCV), or syphilis. Active HBV is defined as Hepatitis B Surface Antigen (HBsAg) or Hepatitis B e Antigen (HBeAg) positivity with HBV DNA≥2000 IU/ml (10⁴ copies/ml). If HBV DNA is below this level, antiviral therapy is required until one year post - study. Active HCV is defined as HCV RNA above the assay's upper limit. For syphilis, a positive non-treponemal test requires confirmation with a treponemal antibody test. If the latter is negative and the investigator confirms past infection with syphilitic cure, the subject can be included;f) Known human immunodeficiency virus （HIV） positivity or primary immunodeficiency;g) Deemed unsuitable for study participation due to a history of psychosis, family history of psychiatric illness, or mood disorders, as determined by the investigator or psychiatrist;h) Uncontrolled hypertension (systolic BP≥180mmHg and/or diastolic BP≥110mmHg);i) Severe medical conditions with a risk of major bleeding or history of major bleeding.
12. Concomitant use of drugs that may prolong the QT interval or cause torsades de pointes.
13. History of alcohol or drug abuse within the past year.
14. Subjects deemed unsuitable for this treatment regimen by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-06-05 (Estimated); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
MTD | Up to 52 weeks
  Maximum Tolerated Dose
DLT | Up to 52 weeks
  Dose-Limiting Toxicity
Proportion of Subjects With Hematocrit (HCT) < 45% | Up to 100 weeks
  The proportion of subjects with HCT<45% following at least 21 days without or with specified therapies (phlebotomy or erythrocytapheresis).

SECONDARY OUTCOMES:
AUC0-∞ | Pre-dose to 168h post-dose on day 1; Pre-dose to 168h post-dose on day 85 (day 85±3 days).
  The area under the plasma concentration-time curve from time zero to infinity.
AUC0-last | Pre-dose to 168h post-dose on day 1; Pre-dose to 168h post-dose on day 85 (day 85±3 days).
  The area under the plasma concentration-time curve from administration to the last measurable concentration time point.
Cmax | Pre-dose to 168h post-dose on day 1; Pre-dose to 168h post-dose on day 85 (day 85±3 days).
  The maximum plasma drug concentration
Tmax | Pre-dose to 168h post-dose on day 1; Pre-dose to 168h post-dose on day 85 (day 85±3 days).
  The time to reach maximum plasma drug concentration
t1/2 | Pre-dose to 168h post-dose on day 1;Pre-dose to 168h post-dose on day 85 (day 85±3 days).
  The time for plasma drug concentration to halve
CL/F | Pre-dose to 168h post-dose on day 1; Pre-dose to 168h post-dose on day 85 (day 85±3 days).
  The ratio of an orally administered drug's absorbed amount to the administered dose
Changes in White Blood Cell (WBC) | Up to 100 weeks
  Changes in WBC over time relative to baseline.
Changes in Platelet (PLT) | Up to 100 weeks
  Changes in PLT over time relative to baseline.
Time to First HCT Response | Up to 100 weeks
  Time to first HCT response (days from study drug administration to HCT <45% without phlebotomy or erythrocytapheresis during this period).
Duration of Peripheral Blood HCT Response | Up to 100 weeks
  Duration of peripheral blood HCT response (days from achieving HCT <45% after study drug administration to HCT ≥45% without phlebotomy or erythrocytapheresis during this period).
Changes in Serum Iron | Up to 100 weeks
  Serum Iron changes at each dose level.
Changes in Hepcidin | Up to 100 weeks
  Hepcidin changes at each dose level.
Changes in Ferritin | Up to 100 weeks
  Ferritin changes at each dose level.
Changes in Transferrin Saturation | Up to 100 weeks
  Transferrin saturation changes at each dose level.
Changes in Spleen Volume Size | Up to 100 weeks
  Mean and percentage changes from baseline in spleen volume.
Symptom Improvement | Up to 100 weeks
  Symptom changes are assessed using the Myeloproliferative Neoplasms 10 (MPN10) questionnaire, with symptoms rated on a scale from 1 to 10 (0 if absent), where 1 indicates the mildest severity and 10 the most severe.
Thrombotic and Hemorrhagic Events | Up to 100 weeks
  The proportion of subjects without thrombotic or hemorrhagic events.
Occurrence of Adverse Events (AEs) | Up to 36 months
  Occurrence of AEs will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events Version 5.0 (NCI CTCAE V5.0).

CONTACTS AND LOCATIONS:
Overall Officials: Zhijian Xiao, Ph.D, Principal Investigator — Blood Diseases Hospital, Chinese Academy of Medical Sciences; Hongyan Tong, Ph.D, Principal Investigator — Zhejiang University
Locations (1):
- Blood Diseases Hospital, Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality, China